CLINICAL TRIAL: NCT02132520
Title: A Brain Centered Neuroengineering Approach for Motor Recovery After Stroke: Combined Repetitive Transcranial Magnetic Stimulation and Brain-Computer Interface Training
Brief Title: A Brain Centered Neuroengineering Approach for Motor Recovery After Stroke: Combined rTMS and BCI Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1306M36401; CBET-1264562 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2014-04-08; First posted 2014-05-07 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Hemiparesis; Stroke
Keywords: Hemiparesis; Stroke; Rehabilitation; Transcranial Magnetic Stimulation, Repetitive; Electroencephalography; Functional Neuroimaging; Brain-Computer Interface
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Subjects receiving standard-of-care physical therapy only.
- Sham rTMS + Real BCI Training (Sham Comparator): Subjects will receive sham rTMS followed by real BCI training.
  Interventions: Device: rTMS; Behavioral: BCI Training
- Real rTMS + Real BCI Training (Active Comparator): Subjects will receive real rTMS followed by real BCI training.
  Interventions: Device: rTMS; Behavioral: BCI Training

INTERVENTIONS:
Device: rTMS — Low frequency rTMS (either real or sham) will be applied to the contralesional hemisphere at a rate of 1Hz for 10 minutes.
  Arms: Real rTMS + Real BCI Training; Sham rTMS + Real BCI Training
Behavioral: BCI Training — BCI training will consist of a series of EEG-based motor-imagery tasks with virtual feedback presented on a computer screen.
  Arms: Real rTMS + Real BCI Training; Sham rTMS + Real BCI Training

SUMMARY:
The purpose of this study is to determine whether the combination of low frequency repetitive transcranial magnetic stimulation (rTMS) and motor-imagery-based brain computer interface (BCI) training is effective for enhancing motor recovery after stroke.

The PI's hypothesis is that, in comparison with traditional physical therapy alone, subjects receiving supplementary rTMS and BCI training will show greater functional improvements in hand motor ability over time as well as recovery of normal motor connectivity patterns.

DETAILED DESCRIPTION:
The goal of the present study is to develop and evaluate a brain based approach to improve motor recovery after stroke, by combining rTMS and BCI training. Treatments will consist of low frequency rTMS applied to the contralesional hemisphere, followed by BCI training to encourage activity within the lesioned hemisphere. The primary objective of this study is to test the main hypothesis above in a stroke patient population. Subjects will also undergo a period of BCI only treatments after completion of the combined rTMS and BCI portion.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Cortical or subcortical stroke with isolated unilateral motor paresis
* At least 3 months but no greater than 12 months post stroke and in stable conditions as judged by patient's physician
* Impaired hand function compared to nonparetic side but at least 10 degrees of active finger extension
* Able to ambulate at least 50 feet with minimal stand-by assistance
* Upper Extremity Fugl Meyer (Fugl-Meyer et al., 1975) score of greater than or equal to 20 out of 66
* Beck Depression Inventory (Beck et al., 1961) less than or equal to 19 out of 63
* Mini-mental State Examination score (Folstein et al., 1975) greater than or equal to 24 out of 30
* Must have an ipsilesional motor-evoked potential (MEP) in response to TMS
* Must be stable outpatients currently undergoing rehabilitation consistent with the current standards of care
* Must be able to communicate clearly in English
* Must be able to provide consent in writing.

Exclusion Criteria:

* Personal history of epilepsy or seizures within the past 2 years
* Previous surgical procedure to the spinal cord
* Any MRI incompatible devices
* Pregnancy
* Claustrophobia
* Breathing disorder
* Hearing problems or ringing in the ears
* Bilateral motor paresis or paralysis or those patients that would require significant medical monitoring or management beyond that of a stable outpatient
* Cognitive deficits, other non-motor neurological impairment, bilateral motor paresis or paralysis or those patients that would require significant medical monitoring or management beyond that of a stable outpatient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
Started | 0 | 1 | 2
Completed | 0 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the control (no real or sham rTMS) group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training | Total
Number analyzed (Participants) | 0 | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] |  | 37 [37 to 37] | 64.5 [60 to 69] | 55.3 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1 | 2
  Male |  | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cortical Excitability and Cortical Activation Patterns as Measured by MRI and Functional MRI
Description: The MRI and functional MRI will evaluate the extent to which cortical areas are recruited both during rest and during movement related tasks. This is quantified by a laterality index, calculated as the ratio of activations of ipsi- and contra-lesional precentral gyri during a paretic hand tracking task. A LI of -1 corresponds to entirely contralesional activation, while a value of +1 corresponds to entirely ipsilesional activation.
Time Frame: Baseline, Post-Test 1 (3 weeks), Post-Test 2 (6 weeks)
Population: The laterality index was not calculated for one subject in post-test 2 as no activation overlapped with the ipsilesional or contralesional precentral gyrus.
Measure: Mean (Full Range); unit: Laterality index
Arm/Group | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
Number analyzed (Participants) | 1 | 2
Laterality index
  Baseline | 0.71 [0.71 to 0.71] | 0.72 [0.44 to 1]
  Post-test 1 | -0.25 [-0.25 to -0.25] | 0.81 [0.61 to 1]
  Post-test 2: number analyzed (Participants) | 1 | 1
  Post-test 2 | 1 [1 to 1] | 0.80 [0.80 to 0.80]

2. Secondary Outcome: Changes in Hand Motor Function as Measured by the Box and Block Test
Description: Performance on the box and block test with the paretic hand, quantified as the number of 2.5 cm^3 cubes grasped, lifted, and released to transfer between compartments correctly within 60 seconds.
Time Frame: Baseline, Post-Test 1 (3 weeks), Post-Test 2 (6 weeks)
Measure: Mean (Full Range); unit: Number of blocks
Arm/Group | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
Number analyzed (Participants) | 1 | 2
Number of blocks
  Baseline | 26.0 [26.0 to 26.0] | 2.67 [0.33 to 5.01]
  Post-test 1 | 32.3 [32.3 to 32.3] | 1.66 [1.0 to 2.33]
  Post-test 2 | 39.4 [39.4 to 39.4] | 2.84 [1.33 to 4.34]

3. Secondary Outcome: Changes in Paretic Hand Motor Function as Measured by the Finger Tracking Test
Description: The finger tracking test evaluates the subject's ability to track an oscillating wave with either their paretic or non-paretic finger. Subjects wore custom electro-goniometer braces on each hand, each of which included a potentiometer signaling extension and flexion of the index finger metacarpophalangeal joint. Subjects were presented with target stimuli with a random sinusoidal waveform and were instructed to move the corresponding index finger to match the target trace as the cursor moved across the screen with constant velocity. Performance was quantified by an accuracy index, calculated using the ratio of the error to the standard deviation of the target, normalized to the range of motion for each subject.
Time Frame: Baseline, Post-Test 1 (3 weeks), Post-Test 2 (6 weeks)
Measure: Mean (Full Range); unit: Accuracy index
Arm/Group | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
Number analyzed (Participants) | 1 | 2
Accuracy index
  Baseline | 0.005 [0.005 to 0.005] | -0.028 [-0.030 to -0.025]
  Post-test 1 | 0.008 [0.008 to 0.008] | -0.011 [-0.018 to -0.004]
  Post-test 2 | 0.009 [0.009 to 0.009] | -0.008 [-0.015 to -0.001]

4. Secondary Outcome: Changes in Inter-hemispheric Inhibition
Description: Inter-hemispheric Inhibition was evaluated using paired-pulse TMS both for the stroke hemisphere to non-stroke hemisphere direction as well as for the non-stroke hemisphere to the stroke hemisphere direction. IHI was measured by applying TMS to identified left and right motor hotspots at 1 mV threshold intensity, or 130% of the RMT if 1 mV threshold could not be identified, with single unilateral pulses and paired bilateral pulses. IHI was quantified by comparing the paired-pulse peak-to-peak motor evoked potential amplitudes to the corresponding single pulse MEP amplitudes for each direction of stimulation (ipsi- to contra-lesional and contra- to ipsi-lesional).
Time Frame: Baseline, Post-Test 1 (3 weeks), Post-Test 2 (6 weeks)
Measure: Mean (Full Range); unit: PP/SP ratio
Arm/Group | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
Number analyzed (Participants) | 1 | 2
PP/SP ratio
  Baseline, ipsi-to-contralesional | 1.28 [1.28 to 1.28] | 0.64 [0.62 to 0.65]
  Baseline, contra-to-ipsilesional | 1.26 [1.26 to 1.26] | 0.42 [0.34 to 0.49]
  Post-test 1, ipsi-to-contralesional | 0.90 [0.90 to 0.90] | 1.41 [0.86 to 1.97]
  Post-test 1, contra-to-ipsilesional | 0.31 [0.31 to 0.31] | 1.62 [1.10 to 2.15]

5. Other Pre Specified Outcome: Subject Report of Symptoms
Description: The subject report of symptoms assesses whether subject experience any adverse effects as a result of participation in the study.
Time Frame: within 12 weeks of participation
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in the Resting Motor Threshold
Description: The resting motor threshold is a measure of cortical excitability, and will be recorded for both the stroke and non-stroke hemispheres.
Time Frame: Baseline, Post-Test 1 (3 weeks), Post-Test 2 (6 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Sham rTMS + Real BCI Training | Real rTMS + Real BCI Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No